CLINICAL TRIAL: NCT05580770
Title: A Phase 1/2a Open-Label, Dose Escalation and Expansion Study to Investigate the Safety, Pharmacokinetics, Pharmacodynamics and Efficacy of Mirdametinib in Combination With BGB-3245 in Patients With Advanced Solid Tumors
Brief Title: Mirdametinib + BGB-3245 in Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of tolerability of Brimarafenib when given in combination of Mirdametinib
Sponsor: SpringWorks Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MEKRAF-AST-101
Record Dates: First submitted 2022-09-22; First posted 2022-10-14 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — mirdametinib

STUDY DESIGN:
Intervention Model Description: The study will be conducted in two sequential parts: Part 1 dose escalation (Phase 1) and Part 2 dose expansion (Phase 2a).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1 Dose Escalation Cohorts Ranging in Dose (Experimental): Participants with an oncogenic mutation or other genomic aberration of the MAPK pathway
  Interventions: Drug: Mirdametinib; Drug: BGB-3245
- Phase 2 Dose Expansion A (Experimental): Participants with cutaneous melanoma harboring NRAS mutations
  Interventions: Drug: Mirdametinib; Drug: BGB-3245
- Phase 2 Dose Expansion B (Experimental): Participants with NSCLC harboring KRAS mutations
  Interventions: Drug: Mirdametinib; Drug: BGB-3245
- Phase 2 Dose Expansion C (Experimental): Participants with NSCLC or cutaneous melanoma harboring BRAF Class II or Class III mutation or BRAF Fusion mutation
  Interventions: Drug: Mirdametinib; Drug: BGB-3245

INTERVENTIONS:
Drug: Mirdametinib — Mirdametinib administered orally
  Other Names: PD-0325901
Drug: BGB-3245 — BGB-3245 administered orally

SUMMARY:
A Phase 1/2a open-label, multicenter, dose escalation and expansion study of mirdametinib in combination with BGB-3245 in adult participants with histologically confirmed, advanced (American Joint Committee on Cancer (AJCC) Stage III or IV) metastatic or unresectable solid cancer that is refractory to or has progressed during or after at least 1 line of appropriate prior systemic anti-cancer therapy including chemotherapy, immunotherapy, or appropriate targeted therapy, or for which there is no treatment available, or prior standard of care therapy was not tolerated.

ELIGIBILITY:
Key Inclusion Criteria:

* Able to provide informed consent
* At least 18 years of age on day of signing ICF
* Advanced, metastatic or unresectable solid cancer that has not responded to or progressed during or after at least 1 line of appropriate therapy or for which there is no treatment available or prior therapy was not tolerated.
* Part 1: oncogenic mutation or other genomic aberration of the MAPK pathway
* Part 2: oncogenic mutation or genomic aberration defined below:

  * Cohort A: cutaneous melanoma harboring NRAS mutations.
  * Cohort B: non-small cell lung cancer (NSCLC) harboring a KRAS mutation.
  * Cohort C: NSCLC or cutaneous melanoma harboring BRAF Class II or Class III mutations or BRAF Fusion mutation.
* Must have archival tumor tissue or agree to a fresh tumor biopsy at screening
* Measurable disease per RECIST 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
* Adequate organ function and no transfusion within 14 days of first dose

Key Exclusion Criteria:

* Central Nervous System metastases, leptomeningeal carcinomatosis or untreated spinal cord compression
* History of glaucoma
* Active parathyroid disorder or history of malignancy associated hypercalcemia
* Clinically significant cardiac disease within the past 6 months of signing ICF
* History of toxicity from another RAF, MEK, ERK inhibitor requiring discontinuation of treatment from these agents
* Severe or uncontrolled systemic disease
* Inability to swallow oral medications
* Clinically significant active infection (HIV, Hepatitis B or Hepatitis C)
* History of or ongoing Immune Thrombocytopenia (ITP), Von Willebrand disease and/or other past or present bleeding disorders
* Underlying medical conditions in investigator's opinion to be unfavorable to be a part of the study
* Major surgical procedure or significant traumatic injury within 4 weeks prior to first dose or anticipates need for major surgery while on study
* Systemic anti-cancer therapy within 2 weeks or 5 half-lives before first dose
* Concomitant systemic or glucocorticoid therapy within 2 weeks before first dose
* Concomitant medicines that are strong CYP3A4 inhibitors or inducers within 2 weeks or 5 half-lives before first dose
* Live vaccine within 4 weeks before first dose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2023-02-03 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events | Up to 24 months
  Safety and tolerability endpoint evaluation via incidence of treatment emergent Adverse Events (TEAEs).
  TEAEs severities will be graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Maximum Tolerated Dose (Part 1 Only) | Up to 18 months
  The maximum tolerated dose (MTD) for mirdametinib and BGB-3245 administered as a combination, if any, will be based on safety and tolerability during the first 28 days of treatment in Cycle 1.
Recommended Phase 2 Dose (Part 1 Only) | Up to 24 months
  The recommended phase 2 dose (RP2D) for mirdametinib and BGB-3245 administered as a combination will be determined based on safety, tolerability, PK, preliminary anti-tumor efficacy, and other available data.
Objective Response Rate (Part 2 Only) | Up to 24 months
  Preliminary anti-tumor efficacy for the RP2D of mirdametinib and BGB-3245 administered as a combination as assessed by Computed Tomography (CT) or Magnetic Resonance Imaging (MRI). Objective Response Rate (ORR) defined as the proportion of participants with complete response (CR) + partial response (PR) using Response Evaluation Criteria in Solid Tumors (RECIST v1.1).

SECONDARY OUTCOMES:
Objective Response Rate (Part 1 Only) | Up to 24 months
  Preliminary anti-tumor efficacy for the RP2D of mirdametinib and BGB-3245 administered as a combination as assessed by CT or MRI. ORR defined as the proportion of participants with CR + PR using RECIST v1.1
Duration of Response Rate | Up to 36 months
  Duration of response rate in participants treated with the combination of mirdametinib and BGB-3245, defined as the time from response (CR + PR using RECIST v1.1) to disease progression and/or death.
Change in plasma concentrations of mirdametinib and BGB-3245 | Up to 24 months
  To determine the PK of mirdametinib and BGB-3245 administered as a combination in the eligible participant population. Plasma concentrations of mirdametinib and BGB-3245 will be measured to evaluate systemic exposures (AUC, Cmax, Ctrough, and other PK parameters as data allow).

CONTACTS AND LOCATIONS:
Locations (8):
- United States (6):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Yale-New Haven Hospital-Yale Cancer Center, New Haven, Connecticut
  - Massachusetts General Hospital, Boston, Massachusetts
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
- Australia (2):
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Calvary Mater Newcastle, Waratah

IPD SHARING:
Plan to Share IPD: No